CLINICAL TRIAL: NCT03418688
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of COR388 in Older Healthy Volunteers and Patients With Alzheimer's Disease
Brief Title: A Multiple Ascending Dose Study of COR388
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cortexyme Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR388-002
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — COR388

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COR388 (Active Comparator): Increasing doses of COR388 will be administered for 10 days in cohorts 1-3 and for 28 days in cohort 4.
  Interventions: Drug: COR388
- Placebo (Placebo Comparator): Matching placebo capsules will be administered for 10 days in cohorts 1-3 and for 28 days in cohort 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: COR388 — COR388 administered for 10 or 28 days.
  Other Names: COR388 HCl
  Arms: COR388
Drug: Placebo — Placebo administered for 10 or 28 days.
  Arms: Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, multiple ascending dose study to assess the safety and tolerability of ascending repeat doses of COR388 HCl in older healthy male and female subjects and a cohort of Alzheimer's disease subjects.

DETAILED DESCRIPTION:
The study will enroll 3 cohorts of 8 healthy subjects ≥55 and ≤80 years of age at the Clinical Pharmacology Unit (CPU) and 1 cohort of 12 AD subjects ≥55 and ≤80 years of age. Subjects in cohorts 1-3 will receive the study drug or placebo for 10 consecutive days while confined to the CPU. AD patients in cohort 4 will receive the study drug or placebo for 28 days as outpatient. Blood samples samples will be collected for pharmacokinetic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥55 years to ≤80 years of age, at the time of consent;
* Males of reproductive potential must agree to use double-barrier contraceptive measures or avoid intercourse from the first dose of study drug through 90 days after the last dose of study drug.
* Females of child-bearing potential must be non-lactating, have negative serum pregnancy test results at Screening and negative urine pregnancy test results at Day -1; agree to use double-barrier or hormonal contraceptive measures or avoid intercourse from Day -10 through 28 days after the last dose of study drug.
* Stable doses of medications used for stable chronic illnesses that are not prohibited by the protocol are allowed as long as the dose has been stable for 30 days prior to Screening, and no changes are expected during participation in the study;
* Body mass index ≥19 kg/m2 to ≤35 kg/m2 at Screening;
* Good general health as determined by medical history, physical examination, laboratory reports, and 12-lead ECG prior to enrollment;
* Non-smoker and non-tobacco user for a minimum of 6 months prior to the first admission and for the duration of the study;
* Able to swallow capsules;
* Fluent in, and able to read and comprehend, the English language;

Cohort 4 Only:

* Must have probable AD according to the NINDS-ADRD criteria; and an MMSE-2 score ≥14 and ≤25;
* Must have moderate to severe periodontitis according to the CDC-AAP criteria as determined by the study dentist during the screening oral examination;
* If applicable, have a primary caregiver willing to accept responsibility for supervising the treatment (eg, administering study drug) and assessing the condition of the subject throughout the study in accordance with all protocol requirements.
* Provide, if mentally competent and willing, written informed consent. If the subject is not able to provide written informed consent, written informed consent must be obtained from a legally authorized representative on the subject's behalf, and verbal assent may be obtained from the subject. In addition, if the subject has a caregiver, the caregiver will be required to provide written informed consent prior to the subject's participation in the study.

Exclusion Criteria:

* History or current evidence of clinically significant arrhythmia, heart failure, or hypotension in the Investigator's judgment;
* History or current evidence of clinically significant liver disease in the Investigator's judgment;
* Evidence of renal insufficiency defined as an estimated glomerular filtration rate <50 mL/min/1.73m2 at Screening;
* Subjects who received any treatment for periodontitis in the last 90 days including systemic or local antibiotics (eg, PerioChip®), scaling, root planing, or other surgical treatments;
* Uncontrolled medical or psychiatric illness, uncontrolled seizure disorder, or history of major stroke;
* Active, or recent history of, systemic infection within 30 days prior to Screening that required treatment with antibiotics for longer than 1 week;
* History or current evidence of psychiatric or emotional problems that would invalidate giving informed consent or limit the ability of the subject to comply with study requirements;
* History of systemic allergic reaction to any drug that is considered significant by the Investigator;
* History of alcohol or drug abuse or dependence within 12 months of Screening, as determined by the Investigator;
* Positive alcohol screen at Screening or on Day -1;
* Positive urine screen for prohibited drugs
* Positive blood screen for human immunodeficiency virus (1 and 2), hepatitis B surface antigen, or hepatitis C virus antibodies at Screening;
* Any conditions that, in the opinion of the Investigator, would make the subject unsuitable for enrollment, could interfere with the subject's participation in or completion of the study, or could interfere with interpretation of study results;
* Abnormal results of screening laboratory tests, ECG, or MRI of the brain deemed clinically significant by the Investigator;
* The use of any prohibited medication that cannot be stopped or replaced safely, based on the judgment of the Investigator; or
* Participation in another investigational new drug research study involving small molecule drugs within 30 days or biological drugs within 60 days prior to the first dose of study drug.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
AUC | Day 1 and Day 10
  Area under the concentration-time curve
Cmax | Day 1 and Day 10
  Maximum observed drug concentration during a dosing interval
Tmax | Day 1 and Day 10
  Time to Cmax

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pacific Research Network, San Diego, California
  - Bioclinica Research, Orlando, Florida
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No